CLINICAL TRIAL: NCT06983249
Title: Rhomboid Intercostal and Subserratus Plane Block Versus Quadratus Lumborum Block in Management of Postoperative Pain After Open Nephrectomy
Acronym: Nephrectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD186/2024
Record Dates: First submitted 2024-11-28; First posted 2025-05-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2024-09

CONDITIONS: Open Nephrectomy Surgery
Keywords: Rhomboid intercostal subserratus
MeSH Terms: interventions — Nephrectomy

STUDY DESIGN:
Intervention Model Description: The eligible patients will be enrolled in this double blinded study and randomly allocated into one of two parrallel equal groups (25 patients in each group) according to sample size by computer generated random number list. The allocation will be concealed, the data will blind to the study group. Two persons should be blinded; the patient and the investigator who will monitor the patients.
  Groups:
  Patients will be assigned randomly into two equal groups:
  Group (A): patients will receive RISS block under ultrasound guide 30 ml bupivacaine 0.25%.
  Group B "Quadratus lumborum block": patients will Receive ultra sound guided Quadratus Lumborum block using 20 ml Bupivacaine 0.25% on operated side.
Who Masked: Participant
Masking Description: The eligible patients will be enrolled in this double blinded study and randomly allocated into one of two parrallel equal groups (25 patients in each group) according to sample size by computer generated random number litst. The allocation will be concealed, the data will blind to the study group. Two persons should be blinded; the patient and the investigator who will monitor the patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lumborum nerve block in nephrectomy (Experimental): Qudaratus lumborum nerve block ultrasound guided in nephrectomy
  Interventions: Procedure: Quadratus lumborum nerve block in nephrectomy
- Rhomboid intercostal and Sub-serratus nerve block in nephrectomy (Experimental): Rhomboid intercostal and subserratus nerve block ultrasound guided
  Interventions: Procedure: Rhomboid intercostal and Sub-serratus nerve block in nephrectomy

INTERVENTIONS:
Procedure: Rhomboid intercostal and Sub-serratus nerve block in nephrectomy — That block was performed when the patient was in the lateral position. A high frequency linear ultrasound transducer was placed longitudinally on the patient's back, just 2 cm medial to the medial scapular border. Then, the probe was slightly rotated to obtain an oblique parasagittal plane. The following landmarks were identified: the trapezius muscle, rhomboid major muscle, intercostal muscles, pleura, and lungs (from superficial to deep in order of appearance). Under ultrasound guidance, a 22 mm gauge spinal needle was directed to the plane by using high frequency ultrasound guidence (Sono SiteTM, Inc., Bothell, WA 98021, USA) between the rhomboid major and the underlying intercostal muscles and 15 ml bupivacaine (0.25%) was delivered into that plane (after repeated negative aspiration of blood), and its spread was manifested by the hydrodissection and widening of the plane visualized by ultrasound
  Other Names: Rhomboid intercostal and subserratus nerve block
  Arms: Rhomboid intercostal and Sub-serratus nerve block in nephrectomy
Procedure: Quadratus lumborum nerve block in nephrectomy — Ultrasound guided posterior quadrates lumborum block was done in lateral decubitus position and linear probe according to the depth was placed in the midaxillary line in the transverse plane immediately above the iliac crest and then it was slided dorsally until the "Shamrock sign" was clearly identified. In "Shamrock sign" The quadratus lumborum (QL) muscle is seen as a superior leaf of the Shamrock at the apex of the transverse process (TP) of L4
  Other Names: QLB
  Arms: Quadratus lumborum nerve block in nephrectomy

SUMMARY:
Rhomboid intercostal block (RIB) and Rhomboid intercostal block with sub-serratus plane block (RISS) are the two types of plane blocks used for postoperative analgesia after abdominal surgeries.

For achieving proper postoperative analgesia, multimodal regimens have been described for patients undergoing abdominal procedures like cholecystectomy. These multimodal regimens could include opioid medications, non-opioid analgesics (e.g., acetaminophen and ketorolac), and regional blocks. These modalities could be used alone or in combination. This prospective randomised controlled trial was performed to analyse the postoperative analgesic effects of ultrasound guided Quadratus lumborum block and RISS block in managing post operative pain in patients undergoing open nephrectomy.

DETAILED DESCRIPTION:
Open nephrectomy is an important surgery in treatment of patients with renal cancer, ultrasound guidance is rapidly becoming the gold standard for regional anesthesia. There is an evidence matched with improving technology to show that the use of ultrasound has significant benefits over conventional techniques, such as nerve stimulation and loss of resistance. The improved safety and efficacy that ultrasound brings to regional anesthesia helped promote its use and realize the benefits that regional anesthesia has over general anesthesia, such as decreased morbidity and mortality, superior post-operative analgesia, cost-effectiveness, decreased postoperative complications and an improved postoperative course .

The Rhomboid intercostal and subserratus plane block (RISS) is a relatively newer block technique described by Elsharkawy et al.

The RISS provides analgesia for the regions supplied by T3 - T6 thoracic nerves, analgesia of the RISS block may be due to two different mechanisms. First, the block mainly affects the thoracic intercostal dorsal rami emerging under the erector spinae muscle at the level of T3-T9, where it is attached to the transverse spinal processes. Second, the injected local anesthetic may extend to the paravertebral space under the erector spinae muscle Quadratus lumborum block (QLB) is a new abdominal truncal block for controlling somatic pain in both the upper and lower abdomen.

Although the concept of the block is similar to that of lateral transverses-abdominis plane block (TAPB), the extent of the effect has been suggested to be greater because the point of injection is more dorsal. Local anesthetics are administered into the space between the quadratus lumborum muscle and the medial layer of the thoracolumbar fascia to achieve QLB, which can spread to the paravertebral space .

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open nephrectomy.
* ASA physical status II, III
* Sex (males and females)
* Age 40-70 years

Exclusion Criteria:

Patient refusal or with difficulties in comprehending visual analogue scale (VAS) pain scores

* Any contraindications for regional anesthesia. (eg: coagulopathy, use of anticoagulants or antiplatelets...)
* Hypersensitivity to local anesthetics.
* Infection near site of injection.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | One year
  Primary outcome:
  Time of first post operative analgesic demand

SECONDARY OUTCOMES:
Secondary outcome | One year
  -Total analgesic requirement with a rescue analgesic (IV fentanyl 0.5 mic\kg) was given if the patient had a VAS of 4 or more over 0-24, 24-48, and 48-72 h after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Compare between RISS nerve block versus QLB nerve block in management of post operative pain after nephrectomy

REFERENCES:
- [Background] Elsharkawy H, Hamadnalla H, Altinpulluk EY, Gabriel RA. Rhomboid intercostal and subserratus plane block -a case series. Korean J Anesthesiol. 2020 Dec;73(6):550-556. doi: 10.4097/kja.19479. Epub 2020 Feb 12. PMID 32046475
- [Background] West D. Evaluation of rhomboid intercostal and subserratus plane block under direct vision for postoperative analgesia in thoracic surgeries: a prospective, randomized controlled trial, thoracic non-oncologic. Eur J Cardiothorac Surg. 2022 Nov 3;62(6):ezac532. doi: 10.1093/ejcts/ezac532. No abstract available. PMID 36367247
- [Background] Kozanhan B, Semerkant T, Esme H, Canitez A, Iyisoy MS. Evaluation of rhomboid intercostal and subserratus plane block under direct vision for postoperative analgesia in thoracic surgeries: a prospective, randomized controlled trial. Eur J Cardiothorac Surg. 2022 Nov 3;62(6):ezac498. doi: 10.1093/ejcts/ezac498. PMID 36218395